CLINICAL TRIAL: NCT06957912
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Quality of Recovery After Major Noncardiac Surgery: A Randomized Trial.
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation and Quality of Recovery After Major Noncardiac Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-066
Record Dates: First submitted 2025-04-23; First posted 2025-05-06 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Vagus Nerve Stimulation; Transcutaneous Electric Nerve Stimulation; Noncardiac Surgery; Quality of Recovery
Keywords: Transcutaneous auricular vagus nerve stimulation; Noncardiac surgery; Quality of recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous auricular vagus nerve stimulation group (Experimental): Transcutaneous auricular vagus nerve stimulation
  Interventions: Device: Transcutaneous auricular vagus nerve stimulation
- Sham stimulation group (Placebo Comparator): Sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous auricular vagus nerve stimulation — Transcutaneous auricular vagus nerve stimulation is performed using earphone-shaped stimulators (tVNS501, Ruishenan Medical Device, Inc. JiangSu, China) on the left tragus areas of the outer ear for a total of 30 min. Using parameters we have identified through systematic review, electrical stimulation (pulse width: 200-300 μs; frequency: 25 Hz; duty cycles: 50%) is initiated at 200% perceptual threshold (PT) which means the minimum amount of electricity required to perceive electrical stimulation on the skin described as a pricking or tingling sensation. All conscious patients will be told they may or may not feel any sensation from the stimulation.
  The stimulation will be performed between 15:00 and 17:00 on the first day before surgery, at least 30 minutes before the start of surgery and between 08:00 and 10:00 on the first to third day after surgery.
  Other Names: taVNS
  Arms: Transcutaneous auricular vagus nerve stimulation group
Device: Sham stimulation — Sham stimulation is performed using earphone-shaped stimulators (tVNS501, Ruishenan Medical Device, Inc. JiangSu, China) on the left tragus areas of the outer ear for a total of 30 min. Using parameters we have identified through systematic review, electrical stimulation (pulse width: 200-300 μs; frequency: 25 Hz; duty cycles: 50%) is initiated at 200% perceptual threshold (PT) which means the minimum amount of electricity required to perceive electrical stimulation on the skin described as a pricking or tingling sensation. And the current will be automatically switched off after 15 s. All conscious patients will be told they may or may not feel any sensation from the stimulation. The stimulation will be performed between 15:00 and 17:00 on the first day before surgery, at least 30 minutes before the start of surgery and between 08:00 and 10:00 on the first to third day after surgery.
  Arms: Sham stimulation group

SUMMARY:
Transcutaneous auricular vagus nerve stimulation (taVNS) is a novel non-invasive neuromodulation technique. Existing evidence suggested that taVNS improves pain management, sleep quality, inflammatory responses, and gastrointestinal recovery after surgery. This study is designed to test the hypothesis that perioperative use of taVNS may improve quality of recovery in patients after major noncardiac surgery.

DETAILED DESCRIPTION:
The evolution of quality improvement initiatives, such as Enhanced Recovery After Surgery (ERAS) protocols, has shifted perioperative management paradigms toward prioritizing patient-centered subjective experiences such as quality of recovery over traditional outcomes such as mortality, morbidity, or physiological parameter recovery. Poor quality of recovery after surgery not only diminishes patient satisfaction but also correlates with increased 30-day postoperative complications, prolonged hospital stays, and elevated medical expenses.

The vagus nerve is a major component of the parasympathetic nervous system and is a critical relay for neuro-metabolic signals between the abdominal viscera and the brain. The ear is the only area where the vagus nerve is distributed on the body surface, and the auricular branch of the vagus nerve can project to nerve centers such as nucleus of solitary tract in the brainstem and the nucleus coeruleus in the midbrain.

Transcutaneous auricular vagus nerve stimulation (taVNS) can stimulate the auricular branch of the vagus nerve through surface electrodes located in the cymba conchae, and thus activate the vagus nerve circuit, regulate the activity of the brainstem, thalamus, and other brain regions, and regulate the related peripheral organs. Available evidences showed that taVNS reduces inflammatory response to surgery through cholinergic anti-inflammatory pathways, improves analgesia by reducing inflammation and activating serotonin and endorphins analgesic pathways, and promotes gastrointestinal function by regulating peristalsis and secretion of the digestive system; it was also found effective in improving sleep quality and relieving anxiolytic and depressive symptoms. The use of taVNS is relative safe; the incidence of adverse event is low and mainly included transient earache, headache, and local tingling, with no causal association to serious adverse events.

The investigators hypothesize that the application of taVNS in patients undergoing major noncardiac surgery may improve early postoperative quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years but <85 years.
2. Scheduled for elective or limited-time noncardiac surgery with expected duration ≥2 hours.

Exclusion Criteria:

1. Lesions or infections of the auricle skin.
2. Recent or long-term use of cholinergic or anticholinergic medications.
3. Neurosurgery.
4. Expected mechanical ventilation with intubation for ≥1 day after surgery.
5. Diagnosed schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis before surgery.
6. Preoperative left ventricular ejection fraction (LVEF) <30%, or those with sick sinus syndrome, sinus bradycardia (heart rate <50 beats per minute), atrioventricular block of grade II or above, or implanted pacemaker.
7. Inability to communicate due to coma, severe dementia, or language barrier before surgery, or unable to cooperate with intervention.
8. American Society of Anesthesiologists physical status grade >IV, or estimated survival <24 hours.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery scores at 24 hours after surgery | At 24 hours after surgery
  Quality of recovery is assessed using the 15-item Quality of Recovery (QoR-15) Scale. The QoR-15 is a valid, reliable, responsive, and simple-to-use measure that can be applied across a broad range of surgical settings. The scale contains 15 questions that measure five dimensions of patient's health, including: physical comfort, emotional state, physical independence, psychological support, and pain, with scores ranging from 0 (the poorest quality of recovery) to 150 (the best quality of recovery).

SECONDARY OUTCOMES:
Quality of recovery scores at 48 and 72 hours after surgery | At 48 and 72 hours after surgery
  Quality of recovery is assessed using the 15-item Quality of Recovery (QoR-15) Scale. The scale contains 15 questions that measure five dimensions of patient's health, including: physical comfort, emotional state, physical independence, psychological support, and pain, with scores ranging from 0 (the poorest quality of recovery) to 150 (the best quality of recovery).
Pain intensity both at rest and with movement after surgery | Up to 3 days after surgery.
  Pain intensity is assessed with a numerical rating scale (NRS, an 11-point scale where 0=no pain and 10=the worst pain) twice daily (8:00-10:00 am, 18:00-20:00 pm) after surgery.
Subjective sleep quality after surgery | Up to 3 days after surgery.
  Subjective sleep quality is assessed with a numerical rating scale (NRS, an 11-point scale where 0=the best sleep and 10=the worst sleep) daily (8:00-10:00 am) after surgery.
Opioid consumption within 3 days after surgery | Up to 3 days after surgery.
  Opioid consumption is converted to intravenous sufentanil equivalent.
Pain intensity and opioid consumption (PIOC) index within 3 days after surgery. | Up to 3 days after surgery.
  Pain intensity is calculated as area under curve (AUC) of NRS pain score within 3 days after surgery. Opioid consumption (OC) within 3 days after surgery is summarized. Pain intensity and opioid consumption (PIOC) index is calculated as: PIOC=[(AUCmean rank - AUCrank)/AUCmean rank] + [(OCmean rank - OCrank)/OCmean rank]. The range of the sum is from -200% to +200%. Values above 0 indicate increased summed AUC and OC in comparison to all patients.

OTHER OUTCOMES:
Heart rate variability (HRV) before and after each intervention. | Up to 3 days after surgery.
  Heart rate (HR) is recorded via electrocardiographic (ECG) monitoring during a 50-min period of each intervention, i.e., a 10-min period before, a 30-min period during, and a 10-min period after (sham) intervention. Heart rate variability is calculated offline from analyses of RR intervals.
Depression after surgery | On the 5th day or before hospital discharge after surgery.
  Beck Depression Inventory-II scale (scores range from 0 to 63, with higher score indicating more severe depression) is used to assess the severity of depression.
Anxiety after surgery | On the 5th day or before hospital discharge after surgery.
  Beck Anxiety Inventory scale (scores range from 0 to 63, with higher score indicating more severe anxiety) is used to assess the severity of anxiety.
Incidence of postoperative nausea and vomiting | Up to 3 days after surgery.
  Occurrence of postoperative nausea and vomiting and use of antiemetic drugs within 3 days after surgery.
Length of stay in postanesthesia care unit (PACU) after surgery. | Up to 2 hours after surgery.
  Time interval from PACU admission to PACU discharge after surgery.
Length of stay in hospital after surgery | Up to 30 days after surgery.
  Length of stay in hospital after surgery.
Time to first flatus and defecation after surgery | Up to 30 days after surgery.
  Time to first flatus and defecation after surgery.
Incidence of postoperative complications | Up to 30 days after surgery.
  Postoperative complications are generally defined as new-onset conditions that have adverse effects on postoperative recovery and require therapeutic interventions.
All-cause mortality after surgery | Up to 30 days after surgery.
  Death within 30 days after surgery from all causes.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ljungqvist O, de Boer HD, Balfour A, Fawcett WJ, Lobo DN, Nelson G, Scott MJ, Wainwright TW, Demartines N. Opportunities and Challenges for the Next Phase of Enhanced Recovery After Surgery: A Review. JAMA Surg. 2021 Aug 1;156(8):775-784. doi: 10.1001/jamasurg.2021.0586. PMID 33881466
- [Background] Wessels E, Perrie H, Scribante J, Jooma Z. Quality of recovery in the perioperative setting: A narrative review. J Clin Anesth. 2022 Jun;78:110685. doi: 10.1016/j.jclinane.2022.110685. Epub 2022 Feb 18. PMID 35190342
- [Background] Campfort M, Cayla C, Lasocki S, Rineau E, Leger M. Early quality of recovery according to QoR-15 score is associated with one-month postoperative complications after elective surgery. J Clin Anesth. 2022 Jun;78:110638. doi: 10.1016/j.jclinane.2021.110638. Epub 2022 Jan 13. PMID 35033845
- [Background] Kleif J, Gogenur I. Severity classification of the quality of recovery-15 score-An observational study. J Surg Res. 2018 May;225:101-107. doi: 10.1016/j.jss.2017.12.040. Epub 2018 Feb 21. PMID 29605019
- [Background] Leger M, Campfort M, Cayla C, Lasocki S, Rineau E. Postoperative quality of recovery measurements as endpoints in comparative anaesthesia studies: a systematic review. Br J Anaesth. 2021 Jun;126(6):e210-e212. doi: 10.1016/j.bja.2021.03.008. Epub 2021 Apr 21. No abstract available. PMID 33892949
- [Background] Myles PS, Boney O, Botti M, Cyna AM, Gan TJ, Jensen MP, Kehlet H, Kurz A, De Oliveira GS Jr, Peyton P, Sessler DI, Tramer MR, Wu CL; StEP-COMPAC Group; Myles P, Grocott M, Biccard B, Blazeby J, Boney O, Chan M, Diouf E, Fleisher L, Kalkman C, Kurz A, Moonesinghe R, Wijeysundera D. Systematic review and consensus definitions for the Standardised Endpoints in Perioperative Medicine (StEP) initiative: patient comfort. Br J Anaesth. 2018 Apr;120(4):705-711. doi: 10.1016/j.bja.2017.12.037. Epub 2018 Feb 2. PMID 29576111
- [Background] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Decarie-Spain L, Hayes AMR, Lauer LT, Kanoski SE. The gut-brain axis and cognitive control: A role for the vagus nerve. Semin Cell Dev Biol. 2024 Mar 15;156:201-209. doi: 10.1016/j.semcdb.2023.02.004. Epub 2023 Feb 16. PMID 36803834
- [Background] Zou N, Zhou Q, Zhang Y, Xin C, Wang Y, Claire-Marie R, Rong P, Gao G, Li S. Transcutaneous auricular vagus nerve stimulation as a novel therapy connecting the central and peripheral systems: a review. Int J Surg. 2024 Aug 1;110(8):4993-5006. doi: 10.1097/JS9.0000000000001592. PMID 38729100
- [Background] Wang Y, Li SY, Wang D, Wu MZ, He JK, Zhang JL, Zhao B, Hou LW, Wang JY, Wang L, Wang YF, Zhang Y, Zhang ZX, Rong PJ. Transcutaneous Auricular Vagus Nerve Stimulation: From Concept to Application. Neurosci Bull. 2021 Jun;37(6):853-862. doi: 10.1007/s12264-020-00619-y. Epub 2020 Dec 23. PMID 33355897
- [Background] Farmer AD, Strzelczyk A, Finisguerra A, Gourine AV, Gharabaghi A, Hasan A, Burger AM, Jaramillo AM, Mertens A, Majid A, Verkuil B, Badran BW, Ventura-Bort C, Gaul C, Beste C, Warren CM, Quintana DS, Hammerer D, Freri E, Frangos E, Tobaldini E, Kaniusas E, Rosenow F, Capone F, Panetsos F, Ackland GL, Kaithwas G, O'Leary GH, Genheimer H, Jacobs HIL, Van Diest I, Schoenen J, Redgrave J, Fang J, Deuchars J, Szeles JC, Thayer JF, More K, Vonck K, Steenbergen L, Vianna LC, McTeague LM, Ludwig M, Veldhuizen MG, De Couck M, Casazza M, Keute M, Bikson M, Andreatta M, D'Agostini M, Weymar M, Betts M, Prigge M, Kaess M, Roden M, Thai M, Schuster NM, Montano N, Hansen N, Kroemer NB, Rong P, Fischer R, Howland RH, Sclocco R, Sellaro R, Garcia RG, Bauer S, Gancheva S, Stavrakis S, Kampusch S, Deuchars SA, Wehner S, Laborde S, Usichenko T, Polak T, Zaehle T, Borges U, Teckentrup V, Jandackova VK, Napadow V, Koenig J. International Consensus Based Review and Recommendations for Minimum Reporting Standards in Research on Transcutaneous Vagus Nerve Stimulation (Version 2020). Front Hum Neurosci. 2021 Mar 23;14:568051. doi: 10.3389/fnhum.2020.568051. eCollection 2020. PMID 33854421
- [Background] Jin H, Li M, Jeong E, Castro-Martinez F, Zuker CS. A body-brain circuit that regulates body inflammatory responses. Nature. 2024 Jun;630(8017):695-703. doi: 10.1038/s41586-024-07469-y. Epub 2024 May 1. PMID 38692285
- [Background] Wu Z, Zhang X, Cai T, Li Y, Guo X, Zhao X, Wu D, Li Z, Zhang L. Transcutaneous auricular vagus nerve stimulation reduces cytokine production in sepsis: An open double-blind, sham-controlled, pilot study. Brain Stimul. 2023 Mar-Apr;16(2):507-514. doi: 10.1016/j.brs.2023.02.008. Epub 2023 Feb 16. PMID 36801260
- [Background] Patel ABU, Bibawy PPWM, Althonayan JIM, Majeed Z, Gan WL, Abbott TEF, Ackland GL. Effect of transauricular nerve stimulation on perioperative pain: a single-blind, analyser-masked, randomised controlled trial. Br J Anaesth. 2023 Apr;130(4):468-476. doi: 10.1016/j.bja.2022.12.025. Epub 2023 Feb 22. PMID 36822987
- [Background] Kaniusas E, Kampusch S, Tittgemeyer M, Panetsos F, Gines RF, Papa M, Kiss A, Podesser B, Cassara AM, Tanghe E, Samoudi AM, Tarnaud T, Joseph W, Marozas V, Lukosevicius A, Istuk N, Sarolic A, Lechner S, Klonowski W, Varoneckas G, Szeles JC. Current Directions in the Auricular Vagus Nerve Stimulation I - A Physiological Perspective. Front Neurosci. 2019 Aug 9;13:854. doi: 10.3389/fnins.2019.00854. eCollection 2019. PMID 31447643
- [Background] Patel ABU, Weber V, Gourine AV, Ackland GL. The potential for autonomic neuromodulation to reduce perioperative complications and pain: a systematic review and meta-analysis. Br J Anaesth. 2022 Jan;128(1):135-149. doi: 10.1016/j.bja.2021.08.037. Epub 2021 Nov 18. PMID 34801224
- [Background] Hong GS, Pintea B, Lingohr P, Coch C, Randau T, Schaefer N, Wehner S, Kalff JC, Pantelis D. Effect of transcutaneous vagus nerve stimulation on muscle activity in the gastrointestinal tract (transVaGa): a prospective clinical trial. Int J Colorectal Dis. 2019 Mar;34(3):417-422. doi: 10.1007/s00384-018-3204-6. Epub 2018 Dec 5. PMID 30519842
- [Background] Ru O, Jin X, Qu L, Long D, Liu M, Cheng L, Jiang Y. Low-intensity transcutaneous auricular vagus nerve stimulation reduces postoperative ileus after laparoscopic radical resection of colorectal cancer: a randomized controlled trial. Minerva Anestesiol. 2023 Mar;89(3):149-156. doi: 10.23736/S0375-9393.22.16735-0. Epub 2022 Nov 3. PMID 36326770
- [Background] Wu Y, Song L, Wang X, Li N, Zhan S, Rong P, Wang Y, Liu A. Transcutaneous Vagus Nerve Stimulation Could Improve the Effective Rate on the Quality of Sleep in the Treatment of Primary Insomnia: A Randomized Control Trial. Brain Sci. 2022 Sep 26;12(10):1296. doi: 10.3390/brainsci12101296. PMID 36291230
- [Background] Wang L, Zhang J, Guo C, He J, Zhang S, Wang Y, Zhao Y, Li L, Wang J, Hou L, Li S, Wang Y, Hao L, Zhao Y, Wu M, Fang J, Rong P. The efficacy and safety of transcutaneous auricular vagus nerve stimulation in patients with mild cognitive impairment: A double blinded randomized clinical trial. Brain Stimul. 2022 Nov-Dec;15(6):1405-1414. doi: 10.1016/j.brs.2022.09.003. Epub 2022 Sep 21. PMID 36150665
- [Background] Hilz MJ. Transcutaneous vagus nerve stimulation - A brief introduction and overview. Auton Neurosci. 2022 Dec;243:103038. doi: 10.1016/j.autneu.2022.103038. Epub 2022 Sep 27. PMID 36201901
- [Background] Myles PS, Myles DB. An Updated Minimal Clinically Important Difference for the QoR-15 Scale. Anesthesiology. 2021 Nov 1;135(5):934-935. doi: 10.1097/ALN.0000000000003977. No abstract available. PMID 34543410
- [Background] Leger M, Perrault T, Pessiot-Royer S, Parot-Schinkel E, Costerousse F, Rineau E, Lasocki S. Opioid-free Anesthesia Protocol on the Early Quality of Recovery after Major Surgery (SOFA Trial): A Randomized Clinical Trial. Anesthesiology. 2024 Apr 1;140(4):679-689. doi: 10.1097/ALN.0000000000004840. PMID 37976460
- [Background] Myles PS, Myles DB, Galagher W, Chew C, MacDonald N, Dennis A. Minimal Clinically Important Difference for Three Quality of Recovery Scales. Anesthesiology. 2016 Jul;125(1):39-45. doi: 10.1097/ALN.0000000000001158. PMID 27159009
- [Background] Kim AY, Marduy A, de Melo PS, Gianlorenco AC, Kim CK, Choi H, Song JJ, Fregni F. Safety of transcutaneous auricular vagus nerve stimulation (taVNS): a systematic review and meta-analysis. Sci Rep. 2022 Dec 21;12(1):22055. doi: 10.1038/s41598-022-25864-1. PMID 36543841
- [Background] Badran BW, Yu AB, Adair D, Mappin G, DeVries WH, Jenkins DD, George MS, Bikson M. Laboratory Administration of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS): Technique, Targeting, and Considerations. J Vis Exp. 2019 Jan 7;(143):10.3791/58984. doi: 10.3791/58984. PMID 30663712
- [Background] Bu XS, Zhang J, Zuo YX. Validation of the Chinese Version of the Quality of Recovery-15 Score and Its Comparison with the Post-Operative Quality Recovery Scale. Patient. 2016 Jun;9(3):251-9. doi: 10.1007/s40271-015-0148-6. PMID 26518201
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Andersen LPK, Gogenur I, Torup H, Rosenberg J, Werner MU. Assessment of Postoperative Analgesic Drug Efficacy: Method of Data Analysis Is Critical. Anesth Analg. 2017 Sep;125(3):1008-1013. doi: 10.1213/ANE.0000000000002007. PMID 28632527